CLINICAL TRIAL: NCT06023680
Title: The Sedentary to Active Rising to Thrive (START) Trial: A Proof-of-Concept Sedentary Behavior Reduction Program
Brief Title: The Sedentary to Active Rising to Thrive (START) Trial
Acronym: START
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00023391; K01AG076967 (NIH)
Record Dates: First submitted 2023-08-29; First posted 2023-09-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Sedentary Time; Frailty
Keywords: Physical Activity; Walking; Older Adults
MeSH Terms: conditions — Sedentary Behavior; Frailty; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous sedentary reduction intervention (Active Comparator): Structured intervention to progressively replace sedentary time with one daily 30-minute light-intensity walking bout
  Interventions: Behavioral: Continuous sedentary reduction intervention
- Bouted sedentary reduction intervention (Active Comparator): Structured intervention to progressively replace sedentary time with three daily 10-minute light-intensity walking bouts
  Interventions: Behavioral: Bouted sedentary reduction intervention

INTERVENTIONS:
Behavioral: Continuous sedentary reduction intervention — During Phase 1, one minute of sedentary time will be replaced with very light to light intensity walking at three different times during the day, every day for 10 days, reaching three separate 10-minute walking intervals (or bouts).
  During Phase 2, the three 10-minute walking bouts will be gradually combined into one 30-minute bout over the course of 20 days.
  Arms: Continuous sedentary reduction intervention
Behavioral: Bouted sedentary reduction intervention — During Phase 1, one minute of sedentary time will be replaced with very light to light intensity walking at three different times during the day, every day for 10 days, reaching three separate 10-minute walking intervals (or bouts).
  During Phase 2, the three 10-minute walking bouts will be maintained over the course of 20 days.
  Arms: Bouted sedentary reduction intervention

SUMMARY:
The goal of this behavioral clinical trial is to compare two different ways of becoming less sedentary and more active in 60 older adults at elevated risk of becoming frail.

The main question this project aims to answer are whether participants in each intervention are able to gradually replace 30 minutes of sedentary (sitting-like) behavior with very light walking over 60 days.

There are other questions this project aims to answer that include:

1. whether it is easier to replace sedentary behavior with one 30-minute walking bout or three 10-minute walking bouts
2. whether becoming less sedentary and more active leads to feeling better, have less stress, pain, and fatigue and have more confidence in becoming more regularly active
3. whether becoming less sedentary and more active leads to better regulation of inflammation and metabolism

Participants will be randomized into one of two sedentary reduction behavior programs; one program that gradually replaces sedentary time with one 30-minute walking bout and the other program that gradually replaces sedentary time with three 10-minute walking bouts in the morning, afternoon, and evening. Researchers will compare both programs to see which one is easier to achieve and maintain over 60 days.

DETAILED DESCRIPTION:
Initiating and maintaining habitual physical activity is difficult for sedentary older adults, particularly those encumbered by health challenges. The 2018 US Physical Activity Guidelines recommends that all adults perform ≥150 minutes/week of physical activity and reduce sedentary behaviors. Yet, traditional approaches to increase physical activity do little to address sedentary behavior reduction, especially for older adults. Lower sedentary behavior is associated with improved biological and psychosocial health-independent of meeting physical activity guidelines. Thus, there remains a critical need to implement and evaluate a structured way to reduce sedentary behavior as a potential pathway for habitual physical activity engagement.

This project aims to test two prescribe-able and feasible strategies to initiate and incorporate sedentary behavior reduction into daily lifestyle with remote monitoring. The interventions are an inexpensive and low burden approach to reduce sedentary behavior and promote habitual physical activity. Moreover, accelerometer-based outcomes of sedentary behavior are novel in intervention settings, particularly when measured in free-living, real-world settings. Lastly, this project directly addresses a gap of successful remotely deployable interventions geared to initiate and build activity into daily life by replacing sedentary time among older adults.

Aim 1. Explore the effectiveness of 2 interventions to reduce sedentary time in pre-frail older adults over 2 months

Hypothesis 1a. Each intervention will reduce objectively measured daily sedentary time from baseline levels over 2 months.

Hypothesis 1b. The continuous intervention will result in more reduction of objectively measured sedentary time than the bouts intervention.

Aim 2. Explore the dose-response relationship between sedentary time changes and patient-reported outcomes that include fatigue, fatigability, anxiety, general and exercise-based self-efficacy, stress, pain, and mood over 2 months

Hypothesis 2: Decreased daily sedentary time over 2 months is associated with decreased fatigue, fatigability, anxiety, stress, and pain, and increased general and exercise-based self-efficacy and mood over 2 months.

Aim 3. Explore the dose-response relationship between sedentary time changes and biomarkers of frailty-related inflammation, including serum interleukin (IL-6) (pg/mL) and tumor necrosis factor (TNF) -alpha receptor 1 (pg/mL) over 2 months

Hypothesis 3. Decreased daily sedentary time is associated with decreased serum (IL-6) and TNF-alpha receptor 1 over 2 months.

Aim 4. Explore the dose-response relationship between changes in sedentary time with biomarkers of glucose and lipid metabolism (glucose, insulin, total cholesterol (TC), low-density lipoprotein cholesterol (LDLC), triglycerides, high-density lipoprotein cholesterol (HDLC)), a cytokine marker related to frailty (Growth/Differentiation Factor-15; (GDF-15), hemoglobin A1C (hbA1c), non-esterified free fatty acid, and untargeted metabolomics-based markers of energy regulation.

Hypothesis 4. Decreased daily sedentary time is associated with decreased levels of blood glucose, insulin, TC, LDLC, triglycerides and increased HDLC, decreased GDF-15, decreased hbA1c, decreased non-esterified free fatty acid, and lower circulating metabolites necessary for energy regulation over 2 months.

Aim 5. Explore the dose-response and diurnal relationships between changes in sedentary time and interstitial glucose continuously monitored over 24 hours for 14 consecutive days using a Libre Pro sensor at baseline and 2 months later

Hypothesis 5. Decreased sedentary time is associated with decreased overall glucose and different time-of-day glucose levels, coefficient of variation, % of time in glucose at various ranges (e.g., ≥200, ≥180, ≥140, 70-180, 70-140, <70, <54 mg/dL), mean daily difference, and mean amplitude of glycemic excursion) over 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥65 years
* Pre-frail defined as having 1-2 of the following criteria:
* Self-reported unintentional weight loss
* Self-reported fatigue
* Self-reported low activity
* Slowness measured during a 4-m walking test
* Weakness measured with grip strength
* Self-reported regular physical activity <20 minutes/day
* Self-reported willingness to work up to walking for 30 minutes/day
* Self-reported ability to find a place to walk for up to 30 minutes/day
* Agree to all study procedures and assessments
* Ability to provide informed consent

Exclusion Criteria:

* Self-reported diabetes
* Self-reported problems related to alcohol or drugs
* Self-reported inability to walk across a room
* Self-reported use of a walker
* Self-reported requirement of medical supervision when engaging in physical activity
* Fallen >2 times in the past month
* Participation in another clinical trial
* Plan to move out of the area within 6 months
* Inability to provide self-transportation to study assessment visits
* Inability to complete a usual-paced 400m walking test within 15 minutes without sitting or the help of another
* Uncontrolled resting hypertension (>160/90 mmHg)
* Cognitive impairment determined using the Montreal Cognitive Assessment Test

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-11-28 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Sedentary Time | Baseline, 2 months
  Sedentary time measured with a wrist worn monitor containing an accelerometer sensor
  This measurement is collected under a 7-day/24-hour wear protocol at baseline and again 2 months afterwards to determine the change in sedentary time before and after either intervention.
Intervention Difference in the Change in Sedentary Time | Baseline, 2 months
  Comparing the 2-month change in sedentary time between the two interventions

SECONDARY OUTCOMES:
Change in Physical Activity Accumulation | Baseline, 2 months
  Physical activity fragmentation (e.g., broken up activity accumulation) wrist worn monitor containing an accelerometer sensor
Change in Walking Ability | Baseline, 2 months
  Ability to walk measured at a usual walking pace for 400m at baseline and 2 months afterwards.
Change in Walking Speed | Baseline, 2 months
  Walking speed measured at a usual walking pace for 4m at baseline and 2 months afterwards.
Change in Fatigue | Baseline, 2 months
  Fatigue measured using a Fatigue Scale questionnaire measured at baseline and 2 months afterwards.
  On the questionnaire, a score can range from 0-13 where higher scores mean higher fatigue.
Change in Fatigability | Baseline, 2 months
  Fatigability measured using a Pittsburgh Fatigability questionnaire measured at baseline and 2 months afterwards.
  On the questionnaire, a score can range from 0-100 where higher scores mean higher fatigability.
Change in Anxiety | Baseline, 2 months
  Anxiety measured using an Anxiety Scale questionnaire measured at baseline and 2 months afterwards.
  On the questionnaire, a score can range from 0-20 where higher scores mean higher anxiety.
Change in General Self Efficacy | Baseline, 2 months
  General Self Efficacy measured using a General Self Efficacy questionnaire measured at baseline and 2 months afterwards
  On the questionnaire, a score can range from 0-50 where higher scores mean higher general self efficacy.
Change in Exercise-based Self Efficacy | Baseline, 2 months
  Exercise-based Self Efficacy measured using an Exercise-based Self Efficacy questionnaire measured at baseline and 2 months afterwards.
  On the questionnaire, a score can range from 0-90 where higher scores mean higher exercise-based self efficacy.
Change in Stress | Baseline, 2 months
  Stress measured using a Perceived Stress Scale questionnaire measured at baseline and 2 months afterwards.
  On the questionnaire, a score can range from 0-70 where higher scores mean higher stress.
Change in Pain | Baseline, 2 months
  Pain measured using a modified version of the McGill pain questionnaire measured at baseline and 2 months afterwards.
  On the questionnaire, a score can range from 0-5 where higher scores mean greater pain.
Change in Mood | Baseline, 2 months
  Mood measured using a Profile of Mood Status questionnaire measured at baseline and 2 months afterwards.
  On the questionnaire, a score can range from 0-20 where higher scores mean greater mood disturbance.
Change in Inflammation | Baseline, 2 months
  Inflammation measured from blood draws quantifying serum IL-6 (pg/mL) and TNF-alpha receptor 1 (pg/mL) at baseline and 2 months afterwards
Change in Blood Glucose | Baseline, 2 months
  Blood glucose measured from blood draws
Change in Insulin | Baseline, 2 months
  Insulin measured from blood draws
Change in Total Cholesterol | Baseline, 2 months
  Total cholesterol measured from blood draws
Change in Low-Density Lipoprotein Cholesterol | Baseline, 2 months
  Low-density lipoprotein cholesterol measured from blood draws
Change in High-Density Lipoprotein Cholesterol | Baseline, 2 months
  High-density lipoprotein cholesterol measured from blood draws
Change in Triglycerides | Baseline, 2 months
  Triglycerides measured from blood draws
Change in Growth/Differentiation Factor-15 | Baseline, 2 months
  Growth/Differentiation Factor-15 measured from blood draws
Change in Metabolites | Baseline, 2 months
  Untargeted metabolomics-based markers of energy regulation measured from blood draws
Change in Hemoglobin A1c | Baseline, 2 months
  Hemoglobin A1c measured from blood draws
Change in Non-Esterified Free Fatty Acid | Baseline, 2 months
  Non-Esterified Free Fatty Acid measured from blood draws
Change in Interstitial Glucose | Baseline, 2 months
  Interstitial glucose measured using a continuous glucose monitor worn 24-hours each day for 14 consecutive days at baseline and 2 months afterwards. Specific measurements include overall glucose and different time-of-day glucose levels, coefficient of variation, % of time in glucose at various ranges (e.g., ≥200, ≥180, ≥140, 70-180, 70-140, <70, <54 mg/dL), mean daily difference, and mean amplitude of glycemic excursion).

CONTACTS AND LOCATIONS:
Overall Officials: Amal Wanigatunga, PhD, Principal Investigator — Johns Hopkins Blomberg School of Public Health
Locations (2):
- United States (2):
  - Johns Hopkins ProHealth, Baltimore, Maryland
  - Bayview Medical Center, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No